CLINICAL TRIAL: NCT05473793
Title: The Impact of a Dried Vegetable on Bowel Function and Gut Microbiota in Subjects With Bowel Function Issues
Brief Title: Impact of a Dried Vegetable on Bowel Function and Gut Microbiota
Acronym: HappYFiber
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Wageningen University (Other)
Collaborators: WholeFiber BV (Unknown); Wageningen University and Research, Laboratory of Microbiology (Unknown); Wageningen University and Research, Division of Human Nutrition & Health (Unknown); Wageningen University and Research (Other)
Responsible Party: Principal Investigator, Edith Feskens, Prof. dr. Edith Feskens, Wageningen University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: NL80274.091.22
Record Dates: First submitted 2022-07-11; First posted 2022-07-26 (Actual); Last update posted 2025-02-25 (Actual); Status verified 2025-02

CONDITIONS: Bowel Function Dissatisfaction
Keywords: bowel function issues; constipation; gut microbiota; fiber intake; vegetable; intrinsic fiber
MeSH Terms: conditions — Constipation

STUDY DESIGN:
Intervention Model Description: A randomized, placebo-controlled, parallel, double-blind trial with three intervention arms and one control (placebo) arm.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Subjects not receiving the intervention product will consume a placebo (rice puff particles). Neither the investigator, nor the participants, nor the outcome assessor will know who received what. No Care Provider is included in this trial.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Highest fiber dose (Experimental): This arm receives the highest dose of the intervention product, which is 15g dried vegetable per day divided into two portions of each 7.5g, which are consumed during the course of the day in the food of choice.
  Interventions: Dietary Supplement: Dried chicory root particles
- Medium fiber dose (Experimental): This arm receives the highest dose of the intervention product, which is 10g dried vegetable per day divided into two portions of each 5.0g, which are consumed during the course of the day in the food of choice.
  Interventions: Dietary Supplement: Dried chicory root particles
- Lowest fiber dose (Experimental): This arm receives the highest dose of the intervention product, which is 5g dried vegetable per day divided into two portions of each 2.5g, which are consumed during the course of the day in the food of choice.
  Interventions: Dietary Supplement: Dried chicory root particles
- Control (Placebo Comparator): This arm is the control arm receiving as placebo rice puff particles each day, whose amount corresponds iso-calorically to the medium fiber dosage (~ 21 kcal/day).
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Dried chicory root particles — The intervention product consists of chicory root that have been sliced and dried and are provided in the form of particles (~3mm).
  Other Names: brand name: WholeFiber™
  Arms: Highest fiber dose; Lowest fiber dose; Medium fiber dose
Other: Placebo — The control arm receives a placebo consisting of rice puff particles.
  Other Names: Rice puff particles
  Arms: Control

SUMMARY:
A randomized, placebo-controlled, parallel, double-blind trial with three intervention arms and a period of four intervention-weeks that assesses the intake of different dosages of a complex fiber product on bowel function via microbiota changes in subjects that are unsatisfied with their current bowel function.

DETAILED DESCRIPTION:
Background: Bowel function issues can have a substantial effect on quality of life. Additional fiber intake might modulate bowel function and gut microbiota, thereby increasing stool frequency and consistency. This could improve defecation ease, feeling of incomplete bowel emptying and bowel function satisfaction. We hypothesize that a dried vegetable, that is naturally high in fiber within plant cells could improve bowel function in subjects with bowel function issues.

Objective: The main objective of the study is to assess whether a dried multifiber vegetable improves bowel function assessed by stool frequency, consistency, defecation ease, feeling of incomplete bowel emptying and satisfaction. Secondary objectives are to assess whether these effects are dose-dependent and associated with the modulation of the gut microbiota and activity. Furthermore, the adaption of bowel function and adaptation of the gut microbiota and activity over time will be analyzed.

Study design: A parallel, randomized, double-blind, placebo-controlled trial of four weeks with one placebo control and three intervention arms that differ in intervention product dose.

Study population: Healthy human volunteers, 20 - 80y old, with bowel function issues reflected in low stool frequency/consistency, difficulty to defecate, and dissatisfaction with their current bowel function.

Intervention: A vegetable product consisting of dried chicory root cubes containing 85% dietary fiber is added to the daily diet. The intervention product is consumed twice daily for four weeks with a maximum dose of 15 g/day. The control (placebo) consists of easily digestible rice puff particles and is consumed in the same manner as the intervention.

Main study parameters/endpoints: Main study outcome are endpoint (week 4) differences from baseline between the highest dose (15 g/day) of the treatment intervention and placebo in bowel function assessed by changes in stool frequency, stool consistency, ease of defecation, incomplete feeling of bowel emptying and bowel function satisfaction. Secondary endpoints are gut microbiota composition and differences in bowel function, quality of life and constipation symptoms assessment between all doses and placebo. Finally, changes over time in gut microbiota and bowel function will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* 20 - 80 years old
* Unsatisfied with bowel functions (self-reported), rated on a visual analogue scale (VAS, 0-10) as less than 6
* Four or less bowel movements per week (low stool frequency) and/or
* Hard, lumpy or solid stools (Bristol stool form 1-4) during 90% of bowel movements (hard to solid consistency)
* Able to read and understand Dutch or English

Exclusion Criteria:

* Having a history of medical or surgical events that may significantly affect the study outcome: e.g., IBS or IBD patients and subjects with medically diagnosed constipation (i.e., constipation related to anatomic, medication-related, or readily identifiable physiological causes.)
* Less than one bowel movement per week during the screening
* Medical drug use:

  * Antibiotic use within 3 months of the study screenings day
  * Chronic use of antacids and PPI's
  * Use of laxatives during the screening
  * Chronic use of blood glucose lowering medication
* Consumption of supplements containing fibres (other than laxatives), pro-/ post-/ synbiotics 1 month before the screening
* Not willing to provide faecal samples
* Unable to comply with proper study procedures
* For women of childbearing age: current or planned pregnancy, lactation
* Known allergic reactions to plants from the Asteraceae (Compositae) family (e.g., lettuce, daisies, sunflowers, artichokes, sage, tarragon, chamomile, chicory etc.)
* Reported unexplained weight loss or weight gain of greater than 5 kg in the month prior to pre-study screening
* Reported slimming or medically prescribed diet
* Reported macrobiotic lifestyle
* Personnel the Division of Human Nutrition & Health or the Laboratory of Microbiology
* Current participation in other medical scientific research
* Not having a general practitioner
* Not willing to be informed about accidental discoveries in relation to the subjects health

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2022-08-22 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Bowel function (differences highest dose vs placebo) - bowel function satisfaction | Change after the intervention of 4 weeks
  Bowel function satisfaction is rated on a five-point scale (from "0-not at all" to "4-extremely").
Bowel function (differences highest dose vs placebo) - ease of defecation | Change after the intervention of 4 weeks
  Ease of defecation is rated on a five-point scale (from "0-not at all" to "4-extremely").
Bowel function (differences highest dose vs placebo) - feeling of incomplete bowel emptying | Change after the intervention of 4 weeks
  Feeling of incomplete bowel emptying is rated on a five-point scale (from "0-not at all" to "4-extremely").
Bowel function (differences highest dose vs placebo) - stool consistency | Change after the intervention of 4 weeks
  Stool consistency is measured using the Bristol Stool Form Scale (7-point scale from 1=hard to 7=diarrhea).
Bowel function (differences highest dose vs placebo) - stool frequency | Change after the intervention of 4 weeks
  Stool frequency is measured by counting number of bowel movements per week.

SECONDARY OUTCOMES:
Fecal gut microbiota (between dose differences) | Change after the intervention of 4 weeks
  Measured in fecal samples using DNA sequencing. Compared between different fiber dosages and placebo.
Fecal gut microbiota activity (between dose differences) | Change after the intervention of 4 weeks
  Fecal gut microbiota activity is determined by measuring microbial metabolites in fecal samples among which fermentation products (short-chain fatty acids) using HPLC. Compared between different fiber dosages and placebo.
Quality of Life (between dose differences) | Change after the intervention of 4 weeks
  Quality of life is measured using the questionnaire Patient Assessment of Constipation - Quality of Life. Compared between different fiber dosages and placebo.
Constipation-related symptoms (between dose differences) | Change after the intervention of 4 weeks
  Constipation symptoms is measured using the questionnaire Patient Assessment of Constipation - Symptoms. Compared between different fiber dosages and placebo.
Bowel function (between dose differences) - bowel function satisfaction | Change after the intervention of 4 weeks
  Bowel function satisfaction is rated on a five-point scale (from "0-not at all" to "4-extremely").
  Compared between different fiber dosages and placebo.
Bowel function (between dose differences) - ease of defecation | Change after the intervention of 4 weeks
  Ease of defecation is rated on a five-point scale (from "0-not at all" to "4-extremely"). Compared between different fiber dosages and placebo.
Bowel function (between dose differences) - feeling of incomplete bowel emptying | Change after the intervention of 4 weeks
  Feeling of incomplete bowel emptying is rated on a five-point scale (from "0-not at all" to "4-extremely"). Compared between different fiber dosages and placebo.
Bowel function (between dose differences) - stool consistency | Change after the intervention of 4 weeks
  Stool consistency is measured using the Bristol Stool Form Scale (7-point scale from 1=hard to 7=diarrhea). Compared between different fiber dosages and placebo.
Bowel function (between dose differences) - stool frequency | Change after the intervention of 4 weeks
  Stool frequency is measured by counting number of bowel movements per week. Compared between different fiber dosages and placebo.

OTHER OUTCOMES:
Bowel function (weekly changes) - bowel function satisfaction | Weekly development for a period of 4 weeks
  Bowel function satisfaction is rated on a five-point scale (from "0-not at all" to "4-extremely"). Compared between different fiber dosages and placebo.
Bowel function (weekly changes) - ease of defecation | Weekly development for a period of 4 weeks
  Ease of defecation is rated on a five-point scale (from "0-not at all" to "4-extremely").
Bowel function (weekly changes) - feeling of incomplete bowel emptying | Weekly development for a period of 4 weeks
  Feeling of incomplete bowel emptying is rated on a five-point scale (from "0-not at all" to "4-extremely").
Bowel function (weekly changes) - stool consistency | Weekly development for a period of 4 weeks
  Stool consistency is measured using the Bristol Stool Form Scale (7-point scale from 1=hard to 7=diarrhea).
Bowel function (weekly changes) - stool frequency | Weekly development for a period of 4 weeks
  Stool frequency is measured by counting number of bowel movements per week.
Fecal gut microbiota (weekly changes) | Weekly development for a period of 4 weeks
  Measured in fecal samples using DNA sequencing.
Fecal gut microbiota activity (weekly changes) | Weekly development for a period of 4 weeks
  Fecal gut microbiota activity is determined by measuring microbial metabolites in fecal samples among which fermentation products (short-chain fatty acids) using HPLC.

CONTACTS AND LOCATIONS:
Locations (1):
- Wageningen University & Research, Division of Human Nutrition & Health, Wageningen, Gelderland, Netherlands

IPD SHARING:
Plan to Share IPD: No
As the data contains sensitive personal information researchers interested in the data can contact the principal investigator.

REFERENCES:
- [Background] Puhlmann ML, de Vos WM. Back to the Roots: Revisiting the Use of the Fiber-Rich Cichorium intybusL. Taproots. Adv Nutr. 2020 Jul 1;11(4):878-889. doi: 10.1093/advances/nmaa025. PMID 32199025
- [Background] Puhlmann ML, Jokela R, van Dongen KCW, Bui TPN, van Hangelbroek RWJ, Smidt H, de Vos WM, Feskens EJM. Dried chicory root improves bowel function, benefits intestinal microbial trophic chains and increases faecal and circulating short chain fatty acids in subjects at risk for type 2 diabetes. Gut Microbiome (Camb). 2022 Apr 28;3:e4. doi: 10.1017/gmb.2022.4. eCollection 2022. PMID 39295776